CLINICAL TRIAL: NCT03046810
Title: Treatment of Incontinence Associated Dermatitis - Automated
Acronym: TRIAD-A
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: SchwabCare (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SC-01
Record Dates: First submitted 2017-02-06; First posted 2017-02-08 (Estimated); Last update posted 2018-05-31 (Actual); Status verified 2018-05

CONDITIONS: Incontinence, Urinary; Dermatitis; Incontinence, Fecal
MeSH Terms: conditions — Urinary Incontinence; Dermatitis; Fecal Incontinence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Wellness toileting system (Experimental): This group will use the wellness toileting system for their perineal hygiene and treatment of dermatitis
  Interventions: Device: Wellness toileting system

INTERVENTIONS:
Device: Wellness toileting system — This group will use the wash, dry, cleanse, and apply zinc oxide barrier spray routinely for all toileting.
  Other Names: SchwabCare Wellness Toileting System

SUMMARY:
Incontinence and the skin irritation (dermatitis) associated with it are common problems. Treatment of dermatitis is effective, but requires effective cleaning and application of a barrier substance to prevent further contact between urine or feces and the skin. Water based cleansing with the addition of a pH balanced cleanser is more effective than standard abrasive cleansing with paper or a cloth, and is better tolerated by those with skin irritation. Zinc oxide based barriers effectively promote healing and prevent further skin damage. Spray forms are less cumbersome and generally preferred, but are difficult to for the patient to apply independently given the challenge of accessing the perineum.

40 patients, recruited from 3 specialty pelvic floor centers and 1 assisted living center will be provided a device that cleans, dries, and applies zinc oxide barrier spray with each use of the toilet. Dermatitis will be evaluated at the beginning of the study, and at weeks 1, 2 and 6 by medical staff using a standard scale (The Kennedy Scale).Quality of life will be measured using a visual analog scale derived from the quality of life in incontinence scale.

The investigators hypothesize that the device will 1) effectively treat incontinence associated dermatitis, 2) prevent recurrence, and 3) be preferred over standard treatment.

DETAILED DESCRIPTION:
Incontinence and incontinence associated dermatitis (IAD) are common problems. A recent CDC study noted that up to 50% of noninstitutionalized patients aged 65 and older experienced episodes of incontinence at least monthly, and that 40% of those with incontinence develop secondary IAD The treatment of IAD is focused on effective cleaning and prevention of further exposure to irritant liquids and solids through barrier creams. Enzymatic washes have proven efficacy over soap and water, and zinc oxide is the standard of care for barrier function. Combined, effective cleansing and barrier use treats IAD in as little as 6 days, and effectively prevents recurrent skin damage. In one study, an effective preventive regimen of regularly applied skin therapy reduced the incidence of IAD in an at risk population from 25% to 5%. The combination of enzymatic skin cleanser and barrier protection is the standard of care for maintenance of skin integrity in patients with chronic urinary and fecal incontinence.

Adherence to prescribed regimens is a major barrier to regular use of substances applied to the perineum. Difficulty in accessing the perineum make adherence challenging to those with both full and limited mobility, often requiring assistance from a caregiver. The associated loss of independence and dignity are major detriments to quality of life. Novel formulations of zinc oxide, using aerosol based spray application, facilitate use and improve patient acceptance. In a 2014 nursing home based industry study, spray based zinc oxide was preferred by 80% of patients and caregivers, and improved treatment and prevention of IAD in 70% of the study participants.

Adequate cleansing and drying prior to the application of barrier products is key to effective prevention of skin breakdown. Water-based cleaning of the perineum after toileting has been demonstrated to improve hygiene over standard mechanical, paper-based cleansing, especially in those with limited mobility or incontinence. Evidence further demonstrates that the addition of pH balanced cleansers, applied without mechanical abrasion from cloths or wipes, advances hygiene and minimizes risk of secondary infection.

Study Aims

The aims of this study are to evaluate the efficacy of an automated delivery system for cleansing the perineum, and applying zinc oxide barrier spray to effectively treat and prevent incontinence associated dermatitis in a population with active or recurrent IAD. Secondary aims will be to assess preference for the automated delivery system over standard wash and manually applied barrier sprays.

ELIGIBILITY:
Inclusion Criteria:

* Ability to give informed consent.
* Active functional urinary or fecal incontinence
* Kennedy Scale Grade >2 with active incontinence associated dermatitis
* Willingness to have device installed in home/care center

Exclusion Criteria:

* Active perineal infection
* Prior pelvic radiation
* Perineal surgery within the prior 6 months
* Known allergy or sensitivity to applied agents
* Treatment for dermatitis within the prior 2 weeks.
* Pre-existing pressure ulcer stage 2-4
* Weight exceeding 300 pounds
* Known allergy or hypersensitivity to cleanser or zinc oxide barrier spray
* Home bathroom needs excessive upgrades, or needs ownership authorization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2017-04-01 (Actual); Primary Completion 2019-07 (Estimated); Study Completion 2019-09 (Estimated)

PRIMARY OUTCOMES:
Treatment of dermatitis | 6 weeks
  Improvement in the Kennedy Score for Dermatitis

SECONDARY OUTCOMES:
Prevention of recurrent dermatitis | 12 weeks
  prevention of recurrent dermatitis by clinical criteria
Improvement in quality of life | 12 weeks
  Assessed by visual analog scale derived from quality of life in incontinence scale

CONTACTS AND LOCATIONS:
Overall Officials: Richard S Tilson, MD MPH, Principal Investigator — Director of Clinical Investigation
Locations (1):
- Skyline Urology, Torrance, California, United States

IPD SHARING:
Plan to Share IPD: No
No plan to share individual participant data at this time